CLINICAL TRIAL: NCT06919653
Title: Promoting Adherence to Chemotherapy Handling Guidelines Among Oncology Nurses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dania Abu-Alhaija, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-0038; K01OH012671 (NIH)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Chemotherapy Exposure; Handling Guidelines; Oncology Nurse; Adherence

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into intervention and control groups. Nurses in the intervention group will receive the WISH intervention (online individualized education and debriefing sessions) and the traditional education typically offered by their institution. Nurses in the control group will receive the traditional education typically offered through their institution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WISH Intervention Group (Experimental): Participants will receive the WISH intervention (education on chemotherapy exposure risks and safe handling guidelines and debriefing sessions on chemotherapy exposure incidents) in addition to the traditional education on chemotherapy safety typically offered by their institution.
  Interventions: Behavioral: The Workplace program to Improve the Safe Handling of hazardous drugs (WISH)
- Control Group (No Intervention): Participants will not receive intervention in this study. They will receive the traditional education on chemotherapy safety typically offered by their institution.

INTERVENTIONS:
Behavioral: The Workplace program to Improve the Safe Handling of hazardous drugs (WISH) — The WISH intervention is targeted to promote the adherence to chemotherapy handling guidelines among oncology nurses. The WISH intervention will include two components 1) an individualized online educational component on chemotherapy exposure and the safe handling guidelines with incorporating novel instructional technology tools and 2) debriefing sessions on the incidents of chemotherapy exposure.
  Arms: WISH Intervention Group

SUMMARY:
Chemotherapy exposure is a serious occupational hazard affecting oncology nurses. Oncology nurses' adherence to chemotherapy handling guidelines is essential to prevent their exposure to chemotherapy. The goal of this research is to develop, validate, and pilot test an intervention "Workplace program to Improve Safe Handling of hazardous drugs" (WISH), to promote adherence to chemotherapy handling guidelines among oncology nurses. The WISH intervention includes two components: an educational component and debriefing sessions on chemotherapy exposure incidents. First, the research team will use a mixed-methods approach to develop an online educational component on chemotherapy safety, establish the content validity of the educational content based on experts' evaluation, and establish the face validity of the educational content by conducting three qualitative focus groups with oncology nurses (n=4-6 nurses per group). Next, the research team will test the feasibility and acceptability of the intervention using a pilot randomized controlled trial with two groups of oncology nurses, an intervention group (n= 30) and a control group (n=30). We will obtain quantitative and qualitative measures of the intervention feasibility and acceptability. The output is an intervention program targeted to train nurses on safe chemotherapy handling guidelines. Findings will be disseminated through peer-reviewed publications and presentations. The intermediate outcome is the adoption of the intervention program by healthcare institutions to train nurses on chemotherapy handling guidelines. The end outcome is promoting adherence to chemotherapy handling guidelines among oncology nurses.

DETAILED DESCRIPTION:
Oncology nurses are at risk for the dangerous health problems of chemotherapy exposure. Chemotherapy exposure is defined as the direct contact with chemotherapy drugs that occurs through skin absorption, hand-to-mouth ingestion, inhalation, and injection with a sharp contaminated object. In order to prevent chemotherapy exposure incidents among nurses, it is important that nurses follow the safe chemotherapy handling guidelines. Unfortunately, the adherence to these guidelines among nurses is lower than the recommended level. The review of the literature reveals the need for an intervention that promotes the adherence to chemotherapy handling guidelines among oncology nurses. The purpose of this study is to develop, validate, and pilot test an intervention to promote adherence to the chemotherapy handling guidelines among oncology nurses.

Specific aim 1: develop and validate an intervention, WISH intervention, to promote greater adherence to safe chemotherapy handling guidelines among oncology nurses. This intervention includes two components 1) an educational component 2) debriefing sessions. In this aim a mixed-method design will be used to: a) Develop an online educational component on chemotherapy exposure and the safe handling guidelines by the study investigators; b) obtain experts evaluation on the content validity of the educational content; c) conduct 3 focus groups with oncology nurses (n=12-18, 4-6 nurses per group) through Zoom to obtain oncology nurses' judgment on the face validity of the educational component (clarity, relevance of the educational material to nurses' responsibilities, usefulness) and to identify other features of the WISH intervention (frequency and duration of the study activities and the type of the debriefing tool). Content analysis methods will be used to analyze the transcripts of the focus groups.

Specific aim 2: test the feasibility and acceptability of the WISH intervention using a pilot randomized controlled trial. This will include two groups of oncology nurses (n=60); an intervention group (n=30), in which nurses will receive the WISH intervention and traditional education on chemotherapy safety by their institution, and a control group (n=30), in which nurses will receive the traditional education on chemotherapy safety by their institution. Sample size was determined by power calculation.

After the informed consent process, participants will take the pretest, then, they will be randomized into control and intervention groups using computer-allocated random numbers. Nurses in the control group will receive the traditional education offered through their institution. Nurses in the intervention group will receive the WISH intervention (online individualized education and debriefing sessions) and the traditional education offered by their institution. Post-tests will be conducted at 6 weeks and 12 weeks after the intervention for both groups using REDCap, a secure web-based application.

Method for sample size calculation:

The target sample size in this study is 60 nurses. This sample size was calculated based on power calculations. With this sample size, this study is powered to detect an effect size at least 0.65 (at power level 80%, α=0.05). This is a feasibility study in which the attrition rate will be determined. Informed by recommendations from previous studies, we will make every effort to retain participants and engage them in all the study activities. Assuming an attrition rate of 10% (54 nurses; 27 in each group), this study will be powered to detect significant differences in the primary outcome (adherence to chemotherapy handling guidelines) with an effect size of at least 0.69 (at power level 80%, α=0.05)

Methods for data analysis:

Feasibility will be measured in terms of the response rate (percent of nurses who responded relative to the number of potential participants who were reached), retention rates (percent of nurse participants who complete the posttests), the time required to reach the target sample size, and the engagement rate (the percent of actual interactions with participants relative to the planned number of interactions). Acceptability will be measured by the Acceptability of Intervention Measure and the adapted measures of ease of use, usefulness, and satisfaction with the study experience, with open-ended comment question. Content analysis method will be used to analyze participants' qualitative feedback on their satisfaction with the study experience.

Descriptive statistics (mean, standard deviation, median, frequencies, percent) will be used to summarize participants' characteristics and other quantitative variables. Sample t-test or Chi square based on the level of measurement will be used to assess if there are significant differences in the demographic, baseline data, and outcome scores between the intervention and control groups. Baseline differences in sample characteristics will be controlled in analysis using ANCOVA.

ELIGIBILITY:
Inclusion Criteria:

* being at least 18 years old
* able to read and speak English
* working as an oncology nurse for at least 3 months
* handling chemotherapy drugs at work

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Nurses' adherence to chemotherapy handling guidelines | Baseline, 6 weeks after the intervention, and 12 weeks after the intervention
  This variable will be measured using Hazardous Drug Handling Questionnaire. The scores reflect the percentage of time nurses adhere to chemotherapy handling guidelines and range between 0%-100%. A higher score indicates greater adherence to chemotherapy handling guidelines.

SECONDARY OUTCOMES:
Nurses' health beliefs regarding chemotherapy exposure | Baseline, 6 weeks after the intervention, and 12 weeks after the intervention
  This variable will be measured using the health beliefs subscales in the Oncology Nurses Health Behaviors Determinants Scale. These subscales are:
  1. Perceived Threat Subscale: range of scores is 5-25, a higher score indicates greater perceived threat of chemotherapy exposure.
  2. Perceived Benefit Subscale: range of scores is 3 -15, a higher score indicates greater perceived benefits of adherence to chemotherapy handling guidelines.
  3. Perceived Barriers Subscale: range of scores is 5-25, a higher score indicates greater perceived barriers of adherence to chemotherapy handling guidelines.
  4. Perceived Self-Efficacy Subscale: range of scores is 6-30, a higher score indicates greater perceived self-confidence to adhere to chemotherapy handling guidelines.
Knowledge on chemotherapy safety | Baseline, 6 weeks after the intervention, and 12 weeks after the intervention
  This variable will be measured using Chemotherapy Safety Knowledge questionnaire. This questionnaire will be developed by the study investigators; development is in progress.

OTHER OUTCOMES:
Study feasibility | Baseline, 6 weeks after the intervention, and 12 weeks after the intervention
  Study feasibility will be measured in terms of the response rate (percent of nurses who responded relative to the number of potential participants who were reached), retention rates (percent of nurse participants who complete the posttests), the time required to reach the target sample size, and the engagement rate (the percent of actual interactions with participants relative to the planned number of interactions).
Intervention acceptability | 6 weeks after the intervention, and 12 weeks after the intervention
  Acceptability will be measured using Acceptability of Intervention Measure (score range is 4-20) and adapted measures of ease of use (score range is 3-15), usefulness (score range is 4-20), and satisfaction with the study experience (score range is 2-10) with an open-ended comment question. Higher scores indicate more positive acceptability of intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data related to intervention pilot testing will be preserved in the University of Cincinnati Scholar@UC repository. This will enable sharing the data publicly for purposes of validating and replicating the study results. Participants will be consented on the public sharing of the de-identified data.